CLINICAL TRIAL: NCT07285005
Title: A Phase 3, Randomized, Parallel, Multicenter, Double-blind, Placebo-controlled Study to Investigate Efficacy and Safety of KP 001 in Patients Aged ≥2 Years With Common Venous Malformations, Common Lymphatic Malformations, or KTS/CLOVES Syndrome
Brief Title: A Study to Investigate Efficacy and Safety of KP-001 Compared With Placebo in Patients Aged ≥2 Years With Common VM, Common LM, or KTS/CLOVES Syndrome
Acronym: S-KY
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Kaken Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KP-001-303; undecided (Registry Identifier: test test test test)
Record Dates: First submitted 2025-11-19; First posted 2025-12-16 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Venous Malformations; Lymphatic Malformations; Klippel-Trenaunay Syndrome; CLOVES Syndrome
MeSH Terms: conditions — Lymphatic Abnormalities; Klippel-Trenaunay-Weber Syndrome; Congenital Lipomatous Overgrowth, Vascular Malformations, and Epidermal Nevi

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- KP-001 (Experimental)
  Interventions: Drug: KP-001; Drug: Placebo
- placebo (Placebo Comparator)
  Interventions: Drug: KP-001; Drug: Placebo

INTERVENTIONS:
Drug: KP-001 — Oral repeated dose 100mg or lower
Drug: Placebo — Oral repeated dose

SUMMARY:
This is a phase 3, double-blind, randomized, placebo-controlled, parallel group, adaptive, multicenter study planned to be conducted at multiple sites in North America, Canada, Taiwan and South Korea.

The purpose of this study is to measure the efficacy and safety of KP-001 compared with placebo in patients aged ≥2 years with common VM, common LM, or KTS/CLOVES syndrome.

An independent data monitoring committee (DMC) will be established to determine whether to discontinue or continue the study. It will also determine the redesign of the number of cases based on the result of the interim analysis.

The study will comprise the following:

* Screening Period: Up to 42 days prior to the first dose of study intervention.
* Treatment Period 1: This is a double-blind period in which KP-001 100 mg (or lower dose depending on their body weight) or placebo will be administered to patients once daily after breakfast until Week 24.
* Treatment Period 2: After 24 weeks of double blind treatment, all patients will switch to the KP-001 open label extension and treated up to Week 52.
* Follow-up Visit: This visit will occur 30 days after the last dose of study intervention, and assessments will be performed per the SoA.
* Discontinuation Visit: Patients who discontinue study intervention will be requested to continue participating in the study and assessments will be performed per the SoA. If the patients request to withdraw from the study, all tests and evaluations when possible will be performed at Discontinuation visit.

DETAILED DESCRIPTION:
Safety and Exploratory Assessments Vital signs (blood pressure, heart rate, respiratory rate, and body temperature) will be monitored at each scheduled visit for safety.

Safety laboratory assessments will include hematology, serum chemistry, coagulation parameters (e.g., PT/INR, aPTT, fibrinogen), and urinalysis.

Coagulation biomarkers other than D-dimer will be collected for exploratory/safety purposes only and will not be included in the reported outcome measures.

Exploratory analyses may include the relationship between changes in Symptom Numeric Rating Scale (NRS) scores and Patient Global Impression of Severity (PGI-S) scores.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 2 years or older at the time of consent or assent.
2. Patients diagnosed with ISSVA classification of common VM, common (cystic) LM (including mixed type consisting mainly of either VM or LM), or KTS/CLOVES syndrome.
3. Patients who cannot be cured by resection, who are difficult to resect based on the assessment of the Investigator, or who are considered refractory to available treatment by the Investigator, or who have a contraindication to available treatment.
4. Patients with at least one target lesion at least 4 cm in the longest diameter.
5. Patients with at least one MRI-volumetric target lesion at screening that is determined to be evaluable by the central imaging evaluator.
6. Patients with symptomatic disease, defined as:

   ・ For patients ≥8 years old: Pain NRS of ≥1 and ≤8 score at the screening visit will be eligible only if their daily pain NRS recorded via ePRO from screening to Day 1 (Week 0) does not show a maximum absolute change of ≥6 points. If patients are taking analgesic medication, there must be no change in the type or dosage of analgesic during the screening period. If patients do not have qualifiable pain, then Fatigue or Bleeding/Oozing NRS of ≥1 and ≤8 score at the screening visit is required. Patients with ≥6 points absolute change in pain NRS are eligible if at least one of either Fatigue OR Bleeding/Oozing NRS is ≥1 and ≤8.
   * For patients ≥3 years old to <8 years old: Wong-Baker FACES pain rating scale equal to or greater than 2 points at screening visit. Patients who are ≥3 years old to <8 years old without qualifiable pain will be recruited providing they have symptomatic disease as judged in the opinion of the Investigator (ie, any visible lesion or lesion affecting activities of daily living), and as far as they meet other inclusion criteria.
   * For patients 2 years old: Symptomatic disease as judged in the opinion of the Investigator (ie, any visible lesion or lesion affecting activities of daily living), and patients will be recruited as far as they meet other inclusion criteria.
7. Patients whose pain from vascular malformations has been stable for at least 30 days prior to screening and, if taking analgesic medication, does not require a change in the type of analgesic medication or its dosage during the screening period.
8. Patients who agree that they or their partner (if either of them is of childbearing potential) will use appropriate contraception (eg, condom and spermicide combination, low-dose pills or other appropriate contraceptive methods, sterilization, intrauterine device) from the time of consent until 90 days after the last dose of study intervention.
9. Patients or their LAR who are able to give age-appropriate informed consent at the time of screening.
10. Patients who are judged by the Investigator to be able to comply with the instructions of the Investigator and the study coordinator regarding the matters specified in the protocol, such as the use of study intervention and concomitant use of prohibited drugs.

Exclusion Criteria:

1. Patients with the following diseases: Simple telangiectatic malformation, lymphangiomatosis, lymphangiectatic malformation associated with Gorham's disease, lymphangiectasia, familial cutaneous mucocutaneous venous malformation, blue rubber ball-like nevus syndrome, M-CM/MCAP, CLAPO syndrome, Proteus syndrome, Parkes Weber syndrome, Sturge-Weber syndrome, Mafucci syndrome, Osler's disease, Cowden's disease, or Adams-Oliver syndrome.
2. Patients with uncontrolled diabetes mellitus (HbA1c ≥ 7.0%) or diseases with abnormal glucose metabolism (glycogenic diseases, galactosemia, primary lactose intolerance, etc).
3. Patients with ischemic heart disease, arrhythmia, or heart failure (NYHA III or IV).
4. Patients with gastrointestinal disorders that affect drug absorption, as determined by the Investigator.
5. Patients with concomitant or pre-existing serious drug hypersensitivity to PI3Kα inhibitors.
6. Patients with allergy history of grade ≥ 3 and/or history of grade ≥ 3 allergic reactions to drug.
7. Patients with known hypersensitivity to quinine.
8. Patients with concomitant or pre-existing alcohol or drug abuse.
9. Patients with ANC of <1.5×10^9/L.
10. Patients with acute or chronic kidney disease and/or dialysis dependence. Patients with screening eGFR <30 mL/min/1.73m^2 using the beside Schwartz equation for patients aged <18 years of age or CKD-EPI formula for >18 years of age will also be excluded.
11. Patients who are judged by the Investigator to have hepatic impairment.
12. Patients with total bilirubin ≥1.5×ULN for age (unless there is a history of Gilbert Syndrome), ALT ≥2×ULN for age, or AST ≥2×ULN for age will be excluded.
13. Patients with target lesion infection that require treatment within 28 days prior to screening.
14. Patients who have undergone invasive treatment, including sclerotherapy or laser therapy, for the target lesion within 84 days prior to screening.
15. Patients who have used other PI3Kα inhibitors or sirolimus within 84 days prior to screening.
16. Patients who have participated in other clinical studies within 90 days prior to the date of consent.
17. Patients who have participated in a clinical study of KP-001 for any period and have received an investigational drug in the past year.
18. Patients wearing orthodontic appliances, cochlear implants, etc, that may affect MRI, or patients in whom MRI is not feasible or, for example, patients who may have a contraindication to sedation and would require sedation in order to have MRI completed.
19. Patients who are unable to take oral medications.
20. Pregnant women, lactating female patients, female patients who may be pregnant, female patients who wish to become pregnant during the study period and up to 90 days after the last dose of study intervention, or male patients who have partners who wish to become pregnant.
21. Patients with any other illness or medical condition who are judged by the Investigator to be inappropriate as patients for this study.
22. Patients who have received or plan to receive live vaccines during the study period.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-02-26 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
The ratio of volume of target lesions based on MRI | pre-does and at 24weeks post-dose
  To confirm the efficacy of KP-001 100 mg or lower based on body weight administered once daily in patients with vascular malformations (common VM, common LM, or KTS/CLOVES syndrome) in reducing volume of target lesions at 24 weeks

SECONDARY OUTCOMES:
Change from baseline in NRS of symptom | Week 20 through Week 24
  To confirm the efficacy of KP-001 100 mg or lower based on body weight administered once daily in patients with vascular malformations (common VM, common LM, or KTS/CLOVES syndrome) on disease specific patient-reported outcomes from Week 20 through Week 24
The ratio of volume of target lesions based on MRI | Pre-does and at 12 and 52 weeks post-dose
  To confirm the efficacy of KP-001 100 mg or lower based on body weight administered once daily in patients with vascular malformations (common VM, common LM, or KTS/CLOVES syndrome) in reducing volume of target lesions at 12 and 52 weeks
The proportion of patients defined as a responder at 12, 24, and 52 weeks | pre-does and at 12, 24 and 52 weeks post-dose
  To confirm the efficacy of KP-001 100 mg or lower based on body weight administered once daily in patients with vascular malformations (common VM, common LM, or KTS/CLOVES syndrome) using response rate based on change in target lesion volume (MRI) at 12, 24, and 52 weeks
Change from baseline of Brief Pain Inventory short form | pre-does and at 4, 12, 24, 36, and 52 weeks post-dose
  To evaluate the efficacy of KP-001 100 mg or lower based on body weight administered once daily in patients with vascular malformations (common VM, common LM, or KTS/CLOVES syndrome) on patient-reported outcomes at 4, 12, 24, 36, and 52 weeks
Change from baseline of PGI-S (Patient Global Impression of Severity and PGI-I (Patient Global Impression of Improvement) | pre-does and at 4, 12, 24, 36, and 52 weeks post-dose
  To evaluate the efficacy of KP-001 100 mg or lower based on body weight administered once daily in patients with vascular malformations (common VM, common LM, or KTS/CLOVES syndrome) on patient-reported outcomes at 4, 12, 24, 36, and 52 weeks
Change from baseline of EQ-5D | pre-does and at 4, 12, 24, 36, and 52 weeks post-dose
  To evaluate the efficacy of KP-001 100 mg or lower based on body weight administered once daily in patients with vascular malformations (common VM, common LM, or KTS/CLOVES syndrome) on patient-reported outcomes at 4, 12, 24, 36, and 52 weeks
Change from baseline of NRS of symptom | pre-does and at 4, 12, 24, 36, and 52 weeks post-dose
  To evaluate the efficacy of KP-001 100 mg or lower based on body weight administered once daily in patients with vascular malformations (common VM, common LM, or KTS/CLOVES syndrome) on patient-reported outcomes at 4, 12, 24, 36, and 52 weeks
Change from baseline of Wong-Baker Faces of symptom | pre-does and at 4, 12, 24, 36, and 52 weeks post-dose
  To evaluate the efficacy of KP-001 100 mg or lower based on body weight administered once daily in patients with vascular malformations (common VM, common LM, or KTS/CLOVES syndrome) on patient-reported outcomes at 4, 12, 24, 36, and 52 weeks
Change from baseline of PedsQL Fatigue Scale | pre-does and at 4, 12, 24, 36, and 52 weeks post-dose
  To evaluate the efficacy of KP-001 100 mg or lower based on body weight administered once daily in patients with vascular malformations (common VM, common LM, or KTS/CLOVES syndrome) on patient-reported outcomes at 4, 12, 24, 36, and 52 weeks
Change from baseline in CGI-S (Clinician Global Impression of Severity) and CGI-I (Clinician Global Impression of Improvemen) at 12, 24, 36, and 52 weeks | pre-does and at 12, 24, 36, and 52 weeks post-dose
  To evaluate the efficacy of KP-001 100 mg or lower based on body weight administered once daily in patients with vascular malformations (common VM, common LM, or KTS/CLOVES syndrome) in improving clinician-reported outcomes at 12, 24, 36, and 52 weeks
The proportion of patients achieving both ≥20% reduction in target lesion volume AND ≥1 score reduction in NRS of symptom | pre-does and at 12, 24 and 52 weeks post-dose
  To confirm the efficacy of KP-001 100 mg or lower based on body weight administered once daily in patients with vascular malformations (common VM, common LM, or KTS/CLOVES syndrome) using response rate based on change in target lesion volume (MRI) AND disease specific patient-reported outcomes at 12, 24, and 52 weeks
Change from baseline in non-target lesions by MRI | pre-does and at 12, 24 and 52 weeks post-dose
  To evaluate the efficacy of KP-001 100 mg or lower based on body weight administered once daily in patients with vascular malformations (common VM, common LM, or KTS/CLOVES syndrome) in changing non-target lesion at 12, 24, and 52 weeks
Presence of new lesions based on MRI | pre-does and at 12, 24 and 52 weeks post-dose
  To evaluate the efficacy of KP-001 100 mg or lower based on body weight administered once daily in patients with vascular malformations (common VM, common LM, or KTS/CLOVES syndrome) in suppressing presence of new lesions at 12, 24, and 52 weeks
Time to relapse | pre-does and at 12, 24 and 52 weeks post-dose
  To evaluate the efficacy of KP-001 100 mg or lower based on body weight administered once daily in patients with vascular malformations (common VM, common LM, or KTS/CLOVES syndrome) at 12, 24, and 52 weeks regarding time to relapse
Time to disease progression | pre-does and at 12, 24 and 52 weeks post-dose
  To evaluate the efficacy of KP-001 100 mg or lower based on body weight administered once daily in patients with vascular malformations (common VM, common LM, or KTS/CLOVES syndrome) at 12, 24, and 52 weeks regarding time to disease progression
Additional treatment for pain related to vascular malformation | Up to 24 weeks post-dose
  To evaluate the efficacy of KP-001 100 mg or lower based on body weight administered once daily in patients with vascular malformations (common VM, common LM, or KTS/CLOVES syndrome) for up to 24 weeks regarding concomitant medication for vascular malformation
Plasma KP-001 concentration data obtained from sparse sampling for population PK analysis | 8weeks, 16weeks, 20weeks and 32 weeks post-dose
  To evaluate the pharmacokinetics of KP-001 100 mg or lower based on body weight administered once daily in patients with vascular malformations (common VM, common LM, or KTS/CLOVES syndrome) following multiple oral doses
Adverse events | up to 52 weeks post-dose
  To determine the safety of KP-001 100 mg or lower based on body weight administered once daily in patients with vascular malformations (common VM, common LM, or KTS/CLOVES syndrome) for up to 52 weeks
Clinical events relevant to the vascular malformations (bleeding, infection, thromboembolism, and others) | up to 52 weeks post-dose
  To determine the safety of KP-001 100 mg or lower based on body weight administered once daily in patients with vascular malformations (common VM, common LM, or KTS/CLOVES syndrome) for up to 52 weeks

OTHER OUTCOMES:
Change in D-dimer From Baseline to Week 24 | up to 52 weeks post-dose
  Serum D-dimer will be measured as a coagulation biomarker of disease activity in patients with vascular malformations. The change from baseline to Week 24 will be evaluated to explore its clinical relevance.